CLINICAL TRIAL: NCT05500820
Title: A Randomized, Double-Blind Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of CIN-107 Following Multiple Oral Doses in Healthy Subjects
Brief Title: Study With CIN-107 Following Multiple Oral Ascending Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-107-111
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
Keywords: pharmacokinetics (PK), metabolism, baxdrostat
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1: 2.5 mg CIN-107 (Experimental): Subjects on a low salt diet
  Interventions: Drug: CIN-107
- Cohort 2: 5.0 mg CIN-107 (Experimental): Subjects on a low salt diet
  Interventions: Drug: CIN-107
- Cohort 3: 1.5 mg CIN-107 (Experimental): Subjects on a normal salt diet
  Interventions: Drug: CIN-107
- Cohort 4: 2.5 mg CIN-107 (Experimental): Subjects on a normal salt diet
  Interventions: Drug: CIN-107
- Cohort 5: 0.5 mg CIN-107 (Experimental): Subjects on a normal salt diet
  Interventions: Drug: CIN-107
- Cohort 1: 2.5 mg matching placebo (Placebo Comparator): Subjects on a low salt diet
  Interventions: Drug: Matching Placebo
- Cohort 2: 5.0 mg matching placebo (Placebo Comparator): Subjects on a low salt diet
  Interventions: Drug: Matching Placebo
- Cohort 3: 1.5 mg matching placebo (Placebo Comparator): Subjects on a normal salt diet
  Interventions: Drug: Matching Placebo
- Cohort 4: 2.5 mg matching placebo (Placebo Comparator): Subjects on a normal salt diet
  Interventions: Drug: Matching Placebo
- Cohort 5: 0.5 mg matching placebo (Placebo Comparator): Subjects on a normal salt diet
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: CIN-107 — A repeat oral dose of CIN-107 once daily for 10 days.
  Other Names: baxdrostat
  Arms: Cohort 1: 2.5 mg CIN-107; Cohort 2: 5.0 mg CIN-107; Cohort 3: 1.5 mg CIN-107; Cohort 4: 2.5 mg CIN-107; Cohort 5: 0.5 mg CIN-107
Drug: Matching Placebo — A repeat oral dose of matching placebo once daily for 10 days.
  Arms: Cohort 1: 2.5 mg matching placebo; Cohort 2: 5.0 mg matching placebo; Cohort 3: 1.5 mg matching placebo; Cohort 4: 2.5 mg matching placebo; Cohort 5: 0.5 mg matching placebo

SUMMARY:
This is a randomized, double-blind, study to assess the safety, tolerability, PK, and PD of multiple oral doses of CIN-107 when administered to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 18 and 55 years, inclusive, in good health based on medical and psychiatric history, physical examination, ECG, orthostatic vital signs, and routine laboratory tests (blood chemistry, hematology, coagulation, and urinalysis).
2. Body mass index (BMI) between 18 and 30 kg/m2, inclusive.
3. Nonsmokers who have not used nicotine-containing products for at least 6 months prior to the Screening Visit.

Exclusion Criteria:

1. Actively participating in an experimental therapy study; received experimental therapy with a small molecule within 30 days of Day 1, or 5 half-lives, whichever is longer; or received experimental therapy with a large molecule within 90 days of Day 1, or 5 half-lives, whichever is longer.
2. A personal or family history of long QT syndrome, Torsades de Pointes, or other complex ventricular arrhythmias, or family history of sudden death.
3. History of, or current, clinically significant arrhythmias as judged by the Investigator, including ventricular tachycardia, ventricular fibrillation, or atrial fibrillation.
4. Prolonged QTcF (>450 msec) based on the average of triplicate ECGs.
5. Seated blood pressure higher than 150/90 mmHg or lower than 90/50 mmHg.
6. Resting heart rate higher than 100 bpm or lower than 50 bpm , sinus node dysfunction, or clinically significant heart block.
7. Temperature (T) greater than 37.6o C (99.68o F, measured orally), and respiration rate less than 12 and greater than 20 breaths/minute.
8. Postural tachycardia (ie >30 bpm upon standing) or orthostatic hypotension (ie, a fall in systolic blood pressure (SBP) of ≥20 mm Hg or DBP of ≥ 10 mm Hg when a person assumes a standing position).
9. Serum potassium > upper limit of normal of the reference range (ULN) and serum sodium < lower limit of normal of the reference range (LLN).
10. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) values > 1.2 ULN.
11. Positive for human immunodeficiency virus (HIV) antibody, hepatitis C virus (HCV) antibody, or Hepatitis B surface antigen (HBsAg).
12. A known history of porphyria, myopathy, or an active liver disease.
13. Positive drug or alcohol test result or a history of alcoholism or drug abuse within 2 years prior to the first dose of study drug as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition: DSM-IV.
14. Typical consumption of ≥14 alcoholic drinks weekly.
15. Surgical procedures within 4 weeks of check-in or planned elective surgery during the study period.
16. Currently undergoing treatment with weight loss medication or prior weight loss surgery (eg, gastric bypass surgery).
17. Pregnant, breastfeeding, or planning to become pregnant during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data and following the first and last doses of CIN-107, as the data permit.
Time to maximum plasma concentration (Tmax) | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data and following the first and last doses of CIN-107, as the data permit.
Area under the curve from time 0 to the time of last quantifiable plasma concentration (AUC[0-last]) | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data following the final dose of CIN-107, as the data permit.
Area under the curve from time 0 to infinity | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data following the final dose of CIN-107, as the data permit.
Area under the curve over a dosing interval (tau) | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data following the final dose of CIN-107, as the data permit.
Area under the plasma concentration-time curve (AUC) from time 0 to 24 hours | up to Day 2
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data and following the first dose of CIN-107, as the data permit.
Percent of AUC extrapolated | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data following the final dose of CIN-107, as the data permit.
Terminal phase elimination half-life | up to Day 15
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data following the final dose of CIN-107, as the data permit.
Apparent plasma clearance | up to Day 15
  This PK parameter will be determined for CIN-107 using plasma concentration data.
Apparent volume of distribution | Up to Day 15
  This PK parameter will be determined for CIN-107 using plasma concentration data.
The cumulative amount of CIN-107 and CIN-107-M excreted in the urine (Ae) | up to Day 15
  This PK parameter will be calculated using the urine concentrations of CIN-107 and its primary metabolite (CIN-107-M)
Renal clearance (CLR Calculated as Ae/AUC) of CIN-107 and CIN-107-M | up to Day 15
  This PK parameter will be calculated using the urine concentrations of CIN-107 and its primary metabolite (CIN-107-M)
Fraction of the dose excreted renally (fe) | up to Day 15
  This PK parameter will be calculated using the urine concentrations of CIN-107
Number of patients experiencing adverse events (AEs) | up to Day 15
Number of patients experiencing adverse drug reactions | up to Day 15
Number of patients experiencing serious adverse events (SAEs) | up to Day 15
Plasma concentration of aldosterone | up to Day 15
Plasma renin activity | up to Day 15
Plasma concentration of cortisol (free and total) | up to Day 15
Plasma concentration of ACTH (Adrenocorticotropic hormone) | up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace Clinical Pharmacology Unit
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Background] Freeman MW, Bond M, Murphy B, Hui J, Isaacsohn J. Results from a phase 1, randomized, double-blind, multiple ascending dose study characterizing the pharmacokinetics and demonstrating the safety and selectivity of the aldosterone synthase inhibitor baxdrostat in healthy volunteers. Hypertens Res. 2023 Jan;46(1):108-118. doi: 10.1038/s41440-022-01070-4. Epub 2022 Oct 20. PMID 36266539
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-111&attachmentIdentifier=5ae8edfe-848e-4a91-ad8a-ff0a5e360aae&fileName=cin-107-111-report-synopsis_Redacted.pdf&versionIdentifier=